CLINICAL TRIAL: NCT01192035
Title: PI or NNRTI as First-line Treatment of HIV in a West African Population With Low Adherence - the PIONA Trial
Brief Title: PI or NNRTI as First-line Treatment of HIV in West Africa - the PIONA Trial
Acronym: PIONA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital Skejby (Other); Bandim Health Project (Other); Ministry of Health, Guinea-Bissau (Unknown); Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11/CNES/2010
Record Dates: First submitted 2010-08-09; First posted 2010-08-31 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2014-11

CONDITIONS: HIV-1
Keywords: Africa, Western; Antiretroviral Therapy, Highly Active
MeSH Terms: interventions — efavirenz; Nevirapine; lopinavir-ritonavir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NNRTI (Active Comparator)
  Interventions: Drug: Efavirenz or Nevirapine
- Protease inhibitor (Active Comparator)
  Interventions: Drug: Ritonavir-boosted lopinavir

INTERVENTIONS:
Drug: Efavirenz or Nevirapine — 2 NRTIs (lamivudine 150 mg "bis in die - twice a day" (BID) and either zidovudine 300 mg BID if hemoglobin is ≥ 8 g/L or stavudine 30 mg BID if hemoglobin is < 8 g/L) and 1 NNRTI (efavirenz 600 mg "omne in die - once daily" (OD) or nevirapine 200 mg OD for the first 2 weeks and after that 200 mg BID). Efavirenz will be used in all male patients according to national HIV guidelines. Pregnant patients and female patients with a child bearing potential will be treated with nevirapine if CD4+ cell count is ≤ 350 cells/mm3 with close monitoring of liver enzymes during the first 12 weeks in patients with CD4+ cell count >250 cells/mm3. Females beyond childbearing age will be treated with efavirenz.
  Other Names: Stocrin; Sustiva; Viramune
  Arms: NNRTI
Drug: Ritonavir-boosted lopinavir — 2 NRTIs (lamivudine 150 mg BID and either zidovudine 300 mg BID if hemoglobin is ≥ 8 g/L or stavudine 30 mg BID if hemoglobin is < 8 g/L) and 1 PI (ritonavir-boosted lopinavir 400/100 mg BID).
  Other Names: Kaletra; Aluvia
  Arms: Protease inhibitor

SUMMARY:
BACKGROUND: Since 1996 the combination of three or more drugs has been the mainstay of human immunodeficiency virus (HIV) treatment. The most important types of drugs are called nucleotide reverse transcriptase inhibitors (NRTIs), non-nucleotide reverse transcriptase inhibitors (NNRTIs) and protease inhibitors (PIs) Response to treatment is measured as increasing CD4+ cell count and decreasing HIV viral load. A major problem is the development of resistance. NNRTIs are recommended as part of first-line treatment of HIV in Africa but many Africans have a slower NNRTI clearance than Caucasians making them more susceptible for development of resistance in case of treatment interruptions. PIs might therefore be a better option in an African setting with low adherence.

AIM: To evaluate two different treatment regimens in HIV-1 infected patients:

A) A NNRTI (efavirenz/nevirapine) based regimen and B) A PI (ritonavir-boosted lopinavir) based regimen with regard to treatment outcomes. HYPOTHESIS: Treatment with a PI will be superior to treatment with a NNRTI due to less development of resistance.

METHODS: Treatment-naïve adult HIV-1 patients enrolled in an existing cohort The West African Retrovirus and Acquired Immune Deficiency (WARAID) cohort in Guinea Bissau with CD4+ cell count ≤ 350 cells/µL and/or clinical signs of immune suppression (World Health Organization (WHO) clinical stage 3 or 4) will be randomised 1:1 to: Treatment A: 2 NRTIs (lamivudine and either zidovudine or stavudine) and 1 NNRTI (efavirenz or nevirapine) or Treatment B: 2 NRTIs (same as in treatment A) and 1 PI (ritonavir-boosted lopinavir). Primary outcome: Viral load suppression <400 copies/ml 12 months after enrolment.

PERSPECTIVES: Guidelines for treatment of HIV in Africa are more or less a copy of the guidelines used in Europe and North America. Genetic differences in pharmacokinetics, more women infected in Africa and difficulties ensuring good adherence mean that results obtained from Caucasian patients are not directly transferrable to African patients. The results of this study will hopefully help guiding the treatment of HIV in Africa in the future. The investigators believe the HIV infected people in West Africa deserve the same evidence-based medicine as in developed countries.

ELIGIBILITY:
Inclusion Criteria:

* Antiretroviral treatment (ART) naïve HIV-1 infected patients. Women receiving ART during pregnancy can be included.
* Age ≥ 18 years
* CD4+ cell count ≤ 350 cells/µL and/or
* Clinical signs of immune suppression (WHO clinical stage 3 or 4) irrespective of CD4+ cell count.

Exclusion Criteria:

* Tuberculosis (TB) treatment with rifampicin at the time of enrolment.
* Co-infection with HIV-2.
* Grade 3 or 4 alanine transaminase (ALAT) elevation (>5 times upper normal limit).
* Patients with cerebral disturbances that complicates the ability to give informed consent or follow the treatment regime.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2011-05; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Fraction of patients with viral load suppression <400 copies/ml | 12 months after enrolment

SECONDARY OUTCOMES:
Fraction of patients with viral load suppression <50 copies/ml | 12 months after enrolment
Increment of CD4+ cell count of at least 100 cells/µL | 12 months after enrolment
Development of ≥1 resistance mutations involving the treatment regimens used in patients with viral load >400 copies/ml | 12 months after enrolment
Frequency of adverse events and severe adverse events | Within 12 months
Compliance. | Within 12 months
  Compliance defined as the actual amount of medicine taken compared to the planned amount for the same treatment period. A pill count is carried out at each visit.
Incidence of tuberculosis. | Within 12 months
Death. | Within 12 months
  Death at 12 month follow-up. Any patient lost to follow-up will be attempted visited at home by a field assistant 1 month after latest visit due. Information on patient death from family or neighbors will be recorded as a mortality event and a verbal autopsy conducted.
Weight | Within 12 months
  Increase in body mass index (BMI) and frequency of severe weight loss (>10% of presumed or measured body weight).
Plasma cytokine levels | Within 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Sanne Jespersen, MD, Principal Investigator — Aarhus University Hospital Skejby; Alex L Laursen, MD, DMSc, Study Director — Aarhus University Hospital Skejby; Lars Oestergaard, Prof MD DMSc, Study Director — Aarhus University Hospital Skejby; Christian Wejse, MD, PhD, Study Chair — Aarhus University Hospital Skejby
Locations (1):
- Centro de Tratamento Ambulatoria do Hospital Nacional Simão Mendes, Bissau, Guinea-Bissau

REFERENCES:
- [Derived] Jespersen S, Honge BL, Krarup H, Medstrand P, Sorensen A, Medina C, Te DDS, Correira FG, Erikstrup C, Ostergaard L, Wejse C, Laursen AL; Bissau HIV Cohort study group. Protease Inhibitors or NNRTIs as First-Line HIV-1 Treatment in West Africa (PIONA): A Randomized Controlled Trial. J Acquir Immune Defic Syndr. 2018 Nov 1;79(3):386-393. doi: 10.1097/QAI.0000000000001820. PMID 30044302